CLINICAL TRIAL: NCT02456974
Title: Antibiotic Dosing in Pediatric Intensive Care
Acronym: ADIC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Hospital, Antwerp (Other); Queen Fabiola Children's University Hospital (HUDERF/UKZKF) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2012/172
Record Dates: First submitted 2015-05-18; First posted 2015-05-29 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pharmacokinetics; Amoxicillin-clavulanate; Piperacillin-tazobactam; Vancomycin; Teicoplanin; Meropenem; Ciprofloxacin; Amikacin
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples Without DNA — blood samples and urine samples (only for ciprofloxacin)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- amoxicillin-clavulanate: Patients receiving amoxicillin-clavulanate as part of routine clinical care.
  Interventions: Procedure: blood sampling in patients receiving amoxicillin-clavulanate as part of routine clinical care
- piperacilline-tazobactam: Patients receiving piperacilline-tazobactam as part of routine clinical care.
  Interventions: Procedure: blood sampling in patients receiving piperacilline-tazobactam as part of routine clinical care.
- vancomycin: Patients receiving vancomycin as part of routine clinical care.
  Interventions: Procedure: blood sampling in patients receiving vancomycin as part of routine clinical care.
- teicoplanin: Patients receiving teicoplanin as part of routine clinical care.
  Interventions: Procedure: blood sampling in patients receiving teicoplanin as part of routine clinical care.
- meropenem: Patients receiving meropenem as part of routine clinical care.
  Interventions: Procedure: blood sampling in patients receiving meropenem as part of routine clinical care.
- ciprofloxacin: Patients receiving ciprofloxacin as part of routine clinical care.
  Interventions: Procedure: blood sampling and urine smapling in patients receiving ciprofloxacin as part of routine clinical care.
- amikacin: Patients receiving amikcain as part of routine clinical care.
  Interventions: Procedure: blood sampling in patients receiving amikacin as part of routine clinical care.

INTERVENTIONS:
Procedure: blood sampling in patients receiving amoxicillin-clavulanate as part of routine clinical care
  Groups: amoxicillin-clavulanate
Procedure: blood sampling in patients receiving piperacilline-tazobactam as part of routine clinical care.
  Groups: piperacilline-tazobactam
Procedure: blood sampling in patients receiving vancomycin as part of routine clinical care.
  Groups: vancomycin
Procedure: blood sampling in patients receiving teicoplanin as part of routine clinical care.
  Groups: teicoplanin
Procedure: blood sampling in patients receiving meropenem as part of routine clinical care.
  Groups: meropenem
Procedure: blood sampling and urine smapling in patients receiving ciprofloxacin as part of routine clinical care.
  Groups: ciprofloxacin
Procedure: blood sampling in patients receiving amikacin as part of routine clinical care.
  Groups: amikacin

SUMMARY:
Pharmacokinetics of antibiotics in critically ill neonates, infants and children

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the pediatric intensive care unit
* patient age/weight : 1,8 kg-15 years
* patient receiving antibiotic treatment (piperacillin-tazobactam, amoxicillin-clavulanate, vancomycin, teicoplanin, meropenem, ciprofloxacin, amikacin) via intermittent infusion regimen or continuous infusion according to institutional treatment guidelines
* intra-arterial or intravenous access other than the drug infusion line available for blood sampling (arterial line is preferred)

Exclusion Criteria:

* no catheter in place for blood sampling
* absence of parental/patient consent
* known hypersensitivity to beta-lactam antibiotics, glycopeptides, fluoroquinolones, aminoglycosides
* extracorporeal circuit (haemodialysis, ECMO, peritoneal dialysis )

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children admitted to a neonatal or pediatric intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2012-05; Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
To investigate if first-dose blood concentrations with maximum antimicrobial activity are achieved with current dosing regimens. | 2 years (expected)
To investigate if steady-state blood concentrations with maximum antimicrobial activity are achieved with current dosing regimens. | 2 years (expected)

SECONDARY OUTCOMES:
To compare measured first-dose blood concentrations with predefined pharmacodynamic targets (Time above MIC) | 2 years (expected)
To compare measured steady-state blood concentrations with predefined pharmacodynamic targets (Time above MIC) | 2 years (expected)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter De Cock, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Hospital Pharmacy, Ghent, Belgium

REFERENCES:
- [Derived] Dhont E, Standing JF, Beel E, Nguyen TVA, Herck I, Peperstraete H, Vandenberghe W, Bove T, Vandekerckhove K, Verougstraete N, Stove V, Vande Walle J, De Paepe P, De Cock PA. Individualised amoxicillin-clavulanate dosing recommendations for critically ill children with augmented clearance after cardiac surgery. Int J Antimicrob Agents. 2025 Aug;66(2):107513. doi: 10.1016/j.ijantimicag.2025.107513. Epub 2025 Apr 15. PMID 40239747
- [Derived] Van Der Heggen T, Dhont E, Willems J, Herck I, Delanghe JR, Stove V, Verstraete AG, Vanhaesebrouck S, De Paepe P, De Cock PAJG. Suboptimal Beta-Lactam Therapy in Critically Ill Children: Risk Factors and Outcome. Pediatr Crit Care Med. 2022 Jul 1;23(7):e309-e318. doi: 10.1097/PCC.0000000000002951. Epub 2022 Apr 15. PMID 35426861
- [Derived] Aulin LBS, De Paepe P, Dhont E, de Jaeger A, Vande Walle J, Vandenberghe W, McWhinney BC, Ungerer JPJ, van Hasselt JGC, De Cock PAJG. Population Pharmacokinetics of Unbound and Total Teicoplanin in Critically Ill Pediatric Patients. Clin Pharmacokinet. 2021 Mar;60(3):353-363. doi: 10.1007/s40262-020-00945-4. Epub 2020 Oct 8. PMID 33030704
- [Derived] De Cock PA, Desmet S, De Jaeger A, Biarent D, Dhont E, Herck I, Vens D, Colman S, Stove V, Commeyne S, Vande Walle J, De Paepe P. Impact of vancomycin protein binding on target attainment in critically ill children: back to the drawing board? J Antimicrob Chemother. 2017 Mar 1;72(3):801-804. doi: 10.1093/jac/dkw495. PMID 27999035
- [Derived] De Cock PA, Standing JF, Barker CI, de Jaeger A, Dhont E, Carlier M, Verstraete AG, Delanghe JR, Robays H, De Paepe P. Augmented renal clearance implies a need for increased amoxicillin-clavulanic acid dosing in critically ill children. Antimicrob Agents Chemother. 2015 Nov;59(11):7027-35. doi: 10.1128/AAC.01368-15. Epub 2015 Sep 8. PMID 26349821